CLINICAL TRIAL: NCT01554436
Title: Neuropsychological and Psychopathological Prognosis Factors of Smoking Cessation
Brief Title: Neuropsychological Prognosis Factors of Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8269; 2008-A00645-50 (Other: ID-RCB)
Record Dates: First submitted 2012-02-24; First posted 2012-03-15 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2012-03

CONDITIONS: Smoking Cessation; Nicotine Dependence
Keywords: Smoking; Neuropsychology; Abstinence; Prognosis; Nicotine Dependence, Cigarettes, with Other Nicotine-induced Disorders
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Smoking | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients in smoking cessation (Experimental): patients in smoking cessation
  Interventions: Behavioral: neuropsychological assessment

INTERVENTIONS:
Behavioral: neuropsychological assessment — The main criterion of evaluation of the smoking abstinence will be made by the measure of the rate of carbon monoxide (CO) in the expired air between the study start and during the study until 6 months after inclusion.
  The secondary criteria of evaluation are criteria of neuropsychological order, namely the performances in the tests listed: result of NART test,Continuous Performance Test (CPT), Trail Making test, Stroop test, Iowa gambling task. (IGT), Hayling test, N back test, fluence verbal test

SUMMARY:
The low overall effectiveness of available smoking cessation treatment so far, indicate the need for new and more efficacious ways to help smokers maintain abstinence. Smokers are a highly heterogeneous population. Identification of individual characteristics that predict success in smoking cessation is highly desirable to allow designing more specific strategies in order to enhance success in quitting tobacco.The main objective of this study is to assess whether the presence of certain neuropsychological deficits found before the initiation of smoking cessation is associated with a greater relapse rate.The secondary objectives concern how neuropsychological performance are involved in motivation and craving in the whole sample of smokers or in subsample. Long-term perspective is to define clinical or neuropsychological factors associated with agood or poor prognosis for success and provived more specific and therefore more effective care.

DETAILED DESCRIPTION:
This is a prospective multicenter study. Patients will be recruited to anti tobacco consultations in the Montpellier and Clermont-Ferrand University Hospitals. The initial assessment includes a clinical assessment of smoking history, Axis I disorders history, motivation to quit and craving, a neuropsychological assessment : NART, RVIP task, trail Making Test, Stroop, Iowa gambling task, Hayling test, N back, verbal fluency. Then patients will be reviewed 3 times in 6 months. These visits include: CO level and cigarette consumption since the last visit, cessation strategy (medication, observance … ), tobacco craving questionnary, withdrawal symptoms, abstinence.

The primary endpoint will be smoking abstinence objectified by the rate of carbon monoxide measured at each visit. Subjects who emerge from the study prematurely, especially patients lost to follow will be considered as failures in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-60 years old
* Patient applying for withdrawal regardless of the number of P / A, the length of smoking.
* Patient with nicotine dependence (Fagerstrom Test score > or = 3)
* Patient able to understand the nature, purpose and methodology of the study
* Patient who gave written informed consent to participate in the study
* Patient agree to cooperate in the clinical and neuropsychological evaluation
* Patient affiliated to a French social security system

Exclusion Criteria:

* Patient with a physical disease being able to interact with the cognitive performances: dysthyroidies, pituitary adenomas, neurodegenerative diseases, Parkinson's disease, neoplastic diseases with intellectual location, the central neurological disorders, the cranial traumas.
* Patient in the incapacity to answer at neuropsychological tests
* Patient who can't go back at visits in 6 months
* Pregnancy women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
neuropsychological test | 6 months
  There primary outcome is to assess if smokers with low attentional level (defined has the median of the sample in Nback and RVIP tasks) are at higher level of relapse at 6 months.

SECONDARY OUTCOMES:
Interactions neuropsychological performance and clinical conditions in patients with psychiatric desease | 6 months
  To study other cognitive performance such as decision making abilities on smoking cessation rates at 6 months. To assess in transversal design the link beetween cognitive functioning and some well known pronostic factors of smoking cessation such as motivation or craving before smoking initiation To study the interaction between neuropsychological performance and clinical conditions that may affect cognitive performance on the rate of abstinence. These tests will be done in subgroups of patients with the characteristic of interest such as a current depressive disorders.
Interactions neuropsychological performance and clinical conditions in patients with hyperactivity disorders | 6 months
  To study other cognitive performance such as decision making abilities on smoking cessation rates at 6 months. To assess in transversal design the link beetween cognitive functioning and some well known pronostic factors of smoking cessation such as motivation or craving before smoking initiation To study the interaction between neuropsychological performance and clinical conditions that may affect cognitive performance on the rate of abstinence. These tests will be done in subgroups of patients with the characteristic of interest such as a current hyperactivity disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Sébastien, MD, Principal Investigator — CHRU de Montpellier
Locations (1):
- CHRU de Montpellier, Montpellier, France

REFERENCES:
- [Derived] Flaudias V, Picot MC, Lopez-Castroman J, Llorca PM, Schmitt A, Perriot J, Georgescu V, Courtet P, Quantin X, Guillaume S. Executive Functions in Tobacco Dependence: Importance of Inhibitory Capacities. PLoS One. 2016 Mar 8;11(3):e0150940. doi: 10.1371/journal.pone.0150940. eCollection 2016. PMID 26953688